CLINICAL TRIAL: NCT02602340
Title: Neurocognitive Predictors of Behavioral Therapy Response in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-006-01
Record Dates: First submitted 2015-10-28; First posted 2015-11-11 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Behavioral Activation therapy (Experimental): Participants will complete 10, 90-minute sessions of Behavioral Activation therapy, conducted using a group format. Each group will include 8-12 participants. Behavioral Activation therapy seeks to target behaviors that might maintain or worsen the depression.
  Interventions: Behavioral: Behavioral Activation therapy

INTERVENTIONS:
Behavioral: Behavioral Activation therapy — Behavioral Activation therapy

SUMMARY:
This project aims to identify brain and behavioral characteristics of individuals experiencing symptoms of depression that will predict the effectiveness of Behavioral Activation Therapy. Brain imaging aspects of the study will use functional magnetic resonance imaging (fMRI) and electroencephalography (EEG). Behavioral assessments will include self-report questionnaires, computer-based and observational tasks, and interviews. Assessments will focus on how individuals process positive information (such as reward) and negative information (such as distressing images), as well as how people make decisions. These assessments will be conducted across 2-3 in-person sessions prior to beginning the treatment, and will be repeated across 2-3 in-person sessions after completing treatment. A blood draw will also be conducted pre- and post- treatment. Behavior Activation therapy will consist of 10, 90-minute weekly therapy sessions conducted in small groups.

DETAILED DESCRIPTION:
Anxiety and mood disorders are the most prevalent class of mental health disorders, with lifetime prevalence estimated at 32% and 18%, respectively. These disorders have tremendous personal and socioeconomic impacts (cost >$1500 per-patient/year) due to days lost at work, increased health care utilization, and increased risk of mortality (e.g. cardiovascular disease). First-line treatments for depression include pharmacologic (e.g. selective serotonin reuptake inhibitors) and psychotherapeutic interventions (e.g. cognitive behavioral therapy and behavioral therapy). While both are superior to placebo treatments, only 40-60% of patients experience significant improvement and 15-25% of responders relapse within one year. Thus, long-lasting improvements are experienced by less than 50% of patients. This ineffectiveness has been moderately associated with symptom severity, illness duration, and comorbidity, but these findings do not provide any strategies for improving treatment effectiveness. The current study will seek to identify behavioral or cognitive-affective predictors that indicate how well a patient is responding to treatment so that interventions can be further individualized to more effectively treat refractory patients.

The aim of this study is to identify whether neural, biological, and behavioral responses related to the arbitration of conflicting avoidance and approach drives can predict behavior therapy response for depressed individuals. This aim will be accomplished using behavioral, functional magnetic resonance imaging (fMRI), and genetic analyses pre and post Behavioral Activation therapy. Research subjects will include treatment-seeking individuals with clinically significant symptoms of unipolar depression. Diagnosis will be assessed using structured clinical interviews. Anxious and depressive symptom severity, personality characteristics, and general functioning will be collected via self-report paper-and-pencil questionnaires. Objective measures of approach, avoidance, and conflict behavioral responses will be collected using computer-administered testing and related neural responsivity will be measured using fMRI. For exploratory aims, a blood draw will be collect pre and post-treatment to examine genetic factors that may predict response to behavior therapy. This research has the potential to identify neural and behavioral approach-avoidance characteristics that can help predict which patients are likely to respond to behavior therapy for depression (i.e., predictors of treatment effectiveness) and reveal targets for future treatment modifications.

Aim 1: Clarify the potential contribution of approach-avoidance behaviors and neural responses to depression symptom severity.

Hypothesis 1.1: Approach-related behaviors and conflict arbitration behavior will explain a significant amount of variance in depressive symptoms, above and beyond avoidance-related behavior.

Hypothesis 1.2: Activations within approach-related (i.e., striatum) and conflict arbitration (i.e., lateral PFC) neural circuitry will explain significant variance in depressive symptom severity above and beyond activations within avoidance-related (i.e., amygdala) neural circuitry. Specifically, the investigators expect increased levels of depression to relate to reduced striatal responsivity.

Aim 2: Identify approach-avoidance behaviors and neural responses that predict the effectiveness of behavioral activation therapy (BA) for depressed subjects.

Hypothesis 2.1: Approach-related behaviors and/or conflict arbitration behavior will help predict treatment response above and beyond avoidance-related behavior and baseline symptom severity. Specifically, the investigators expect that decreased reward sensitivity will predict nonresponse of depressed patients to BA.

Hypothesis 2.2: Approach-related and conflict arbitration neural circuitry will help to predict treatment response above and beyond activations within avoidance-related neural circuitry. Specifically, the investigators expect striatal responsivity to reward to predict response of depressed patients to BA.

Aim 3: Identify whether functional improvement with BA is associated with change in approach-avoidance behaviors and/or neural responses.

Hypothesis 3.1: The level of change in reward sensitivity will positively relate to the level of improvement in overall functioning with BA.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-55
2. All genders
3. All races
4. Eligibility as clinically significant depression will be determined by:

   * Scoring greater than 9 on the Patient Health Questionnaire (PHQ-9) or meeting diagnostic criteria for Diagnostic and Statistical Manual (DSM-5) Major Depressive Disorder
   * Self-report that they are interested in obtaining treatment for depression.
   * Through structured diagnostic interviews, it is determined that depressive symptoms are the primary disorder of concern.
5. Able to provide written, informed consent
6. Have sufficient proficiency in English language to understand and complete interviews, questionnaires, and all other study procedures

Exclusion Criteria:

1. Has a history of unstable liver or renal insufficiency; glaucoma; significant and unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, or metabolic disturbance; or any other condition that, in the opinion of the investigator, would make participation not be in the best interest (e.g., compromise the well-being) of the subject or that could prevent, limit, or confound the protocol-specified assessments.
2. A history of drug abuse in the past 6 months, including alcohol, cocaine, marijuana, opiates, amphetamines, methamphetamines, phencyclidine, benzodiazepines, barbiturates, methadone, and oxycodone. Current alcohol use will be ruled out using a breath test and urine testing will be used to rule out current use of other drugs of abuse.
3. Has any of the following Diagnostic and Statistical Manual (DSM-5) disorders:

   * Schizophrenia Spectrum and Other Psychotic Disorders
   * Bipolar and Related Disorders
   * Obsessive-Compulsive and Related Disorders
   * Anorexia or Bulimia Nervosa
   * Substance use disorder within 6 months
4. Moderate to severe traumatic brain injury (>30 min. loss of consciousness or >24 hours posttraumatic amnesia) or other neurocognitive disorder with evidence of neurological deficits, neurological disorders, or severe or unstable medical conditions that might be compromised by participation in the study.
5. Active suicidal ideation with intent or plan
6. Current use of a medication that could affect brain functioning (e.g., anxiolytics, antipsychotics, or mood stabilizers). However, participants reporting current use of prescribed antidepressants (selective serotonin reuptake inhibitors) will be included as long as the dose has been stable for 6 weeks prior to enrolling in the study.
7. Prescription of a medication outside of the accepted range, as determined by the best clinical practices and current research
8. Taking drugs that affect the fMRI hemodynamic response (e.g., methylphenidate, acetazolamide, excessive caffeine intake > 1000 mg/day).
9. MRI contraindications including: cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, shunt (ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators (TENS unit), persons who have ever been a professional metal worker/welder, history of eye surgery/eyes washed out because of metal, vision problems uncorrectable with lenses, inability to lie still on one's back for 60-120 minutes; prior neurosurgery; tattoos or cosmetic makeup with metal dyes, unwillingness to remove body piercings, and pregnancy
10. Unwillingness or inability to complete any of the major aspects of the study protocol, including magnetic resonance imaging (i.e., due to claustrophobia), blood draws, or behavioral assessment. However, failing to complete some individual aspects of these assessment sessions will be acceptable (i.e., being unwilling to answer individual items on some questionnaires or being unwilling to complete a behavioral task).
11. Non-correctable vision or hearing problems

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2015-10-06 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms as measured by the Patient Reported Outcomes Measurement Information System (PROMIS) Depression Scale. | Trajectory of change from pre- to post- treatment; last time point assessed within 6 weeks following last treatment session, on average at 16 weeks after baseline assessment
  Test the predictive effects of imaging and behavioral factors on change in symptoms at baseline compared to within 6 weeks after completing treatment.

SECONDARY OUTCOMES:
Change in depression-related behaviors as assessed by the Behavioral Activation Depression Scale (BADS) Short Form. | Trajectory of change from pre- to post- treatment; last time point assessed within 6 weeks following last treatment session, on average at 16 weeks after baseline assessment
  Test the predictive effects of imaging and behavioral factors on change in symptoms at baseline compared to within 6 weeks after completing treatment.
Change in anxiety symptoms as measured by the Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety Scale. | Trajectory of change from pre- to post- treatment; last time point assessed within 6 weeks following last treatment session, on average at 16 weeks after baseline assessment
  Test the predictive effects of imaging and behavioral factors on change in symptoms at baseline compared to within 6 weeks after completing treatment.
Change in level of disability as measured by the Sheehan Disability Scale | Trajectory of change from pre- to post- treatment; last time point assessed within 6 weeks following last treatment session, on average at 16 weeks after baseline assessment
  Test the predictive effects of imaging and behavioral factors on change in symptoms at baseline compared to within 6 weeks after completing treatment.
Change in depressive symptoms as measured by the Beck Depression Inventory - II. | Change from pre- to post- treatment; last time point assessed within 6 weeks following last treatment session, on average at 16 weeks after baseline assessment
  Test the predictive effects of imaging and behavioral factors on change in symptoms at baseline compared to within 6 weeks after completing treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Robin L Aupperle, Ph.D., Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hollon SD, Stewart MO, Strunk D. Enduring effects for cognitive behavior therapy in the treatment of depression and anxiety. Annu Rev Psychol. 2006;57:285-315. doi: 10.1146/annurev.psych.57.102904.190044. PMID 16318597
- [Background] Hans E, Hiller W. Effectiveness of and dropout from outpatient cognitive behavioral therapy for adult unipolar depression: a meta-analysis of nonrandomized effectiveness studies. J Consult Clin Psychol. 2013 Feb;81(1):75-88. doi: 10.1037/a0031080. PMID 23379264
- [Background] Drevets WC. Neuroimaging and neuropathological studies of depression: implications for the cognitive-emotional features of mood disorders. Curr Opin Neurobiol. 2001 Apr;11(2):240-9. doi: 10.1016/s0959-4388(00)00203-8. PMID 11301246
- [Background] Siegle GJ, Thompson WK, Collier A, Berman SR, Feldmiller J, Thase ME, Friedman ES. Toward clinically useful neuroimaging in depression treatment: prognostic utility of subgenual cingulate activity for determining depression outcome in cognitive therapy across studies, scanners, and patient characteristics. Arch Gen Psychiatry. 2012 Sep;69(9):913-24. doi: 10.1001/archgenpsychiatry.2012.65. PMID 22945620
- [Background] Aupperle RL, Melrose AJ, Francisco A, Paulus MP, Stein MB. Neural substrates of approach-avoidance conflict decision-making. Hum Brain Mapp. 2015 Feb;36(2):449-62. doi: 10.1002/hbm.22639. Epub 2014 Sep 15. PMID 25224633
- [Background] Aupperle RL, Sullivan S, Melrose AJ, Paulus MP, Stein MB. A reverse translational approach to quantify approach-avoidance conflict in humans. Behav Brain Res. 2011 Dec 1;225(2):455-63. doi: 10.1016/j.bbr.2011.08.003. Epub 2011 Aug 6. PMID 21843556
- [Background] Addis, M. and C. Martell, Overcoming Depression One Step at a Time: The New Behavioral Activation Approach to Getting Your Life Back. 2004, Oakland, CA: New Harbinger Publications.
- [Background] Martell, C.R., S. Dimidjian, and R. Herman-Dunn, Behavioral activation for depression: A clinician's guide. 2013: Guilford Press.
- [Background] Dobson KS, Hollon SD, Dimidjian S, Schmaling KB, Kohlenberg RJ, Gallop RJ, Rizvi SL, Gollan JK, Dunner DL, Jacobson NS. Randomized trial of behavioral activation, cognitive therapy, and antidepressant medication in the prevention of relapse and recurrence in major depression. J Consult Clin Psychol. 2008 Jun;76(3):468-77. doi: 10.1037/0022-006X.76.3.468. PMID 18540740